CLINICAL TRIAL: NCT03740828
Title: KIDScore D3 Clinical Study
Status: Completed | Type: Observational
Sponsor: Vitrolife (Industry)
Responsible Party: Sponsor
Other Study IDs: FU1028_Clinical study
Record Dates: First submitted 2018-11-05; First posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Infertility
Keywords: In vitro fertilization; Time-lapse; Assisted Reproduction
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Women undergoing IVF treatment: Device: KIDScore D3 study
  Interventions: Device: KIDScore D3

INTERVENTIONS:
Device: KIDScore D3 — Embryos are scored using the KIDScore D3 algorithm based on annotated morphokinetic parameters.

SUMMARY:
The aim of this study is to demonstrate that the KIDScore D3 may be used to identify those embryos on Day 3 that are most likely to form blastocysts.

DETAILED DESCRIPTION:
The safety and effectiveness of the KIDScore D3 was investigated in a prospective study. The study was performed as a single arm, multicenter clinical study conducted at six sites in the United States. This was a non-interventional clinical study where the KIDScore D3 was not used during patient treatment. Briefly, the purpose of the study was to collect data to evaluate the safety and effectiveness of the KIDScore D3's ability to predict which embryos are most likely to develop to blastocyst stage. This was evaluated by using the KIDScore D3 as adjunct information to traditional morphological grading. Imaging data was collected on embryos cultured to day 5. Embryologists were masked to imaging data and evaluation was only based on morphology and KIDScore D3 scores.

This study aims at analyzing the utilization of established morphology methods with adjunct outcome of an algorithm (KIDScore D3) that provides a score (1 - 5) from timings of morphokinetic events.

A double-blinded, multi-center study, designed to evaluate the odds ratios and other measures for outcomes of methodologies used for embryo assessment: day 3 morphology alone and day 3 morphology with KIDScore D3 results as adjunct information.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing IVF treatment

Exclusion Criteria:

* Less than 5 actively dividing embryos

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women undergoing IVF treatment
Study Population: European women undergoing IVF treatment and imaging of their embryos with the EmbryoScope system
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2017-10-12 (Actual); Study Completion 2017-10-12 (Actual)

PRIMARY OUTCOMES:
Prediction of blastocyst outcome | 1-2 months
  The primary endpoint of this study was to assess the association between the adjunct prediction using KIDScore D3 of blastocyst outcome and the actual blastocyst outcome. The Odds Ratio (OR) for the adjunct prediction of blastulation is required to be statistically significantly greater than 1, for good/fair embryos. This will demonstrate that adjunctive use of KIDScore D3 leads to embryologist predictions for Day 5 blastulation that is informative for blastocysts outcome.

SECONDARY OUTCOMES:
Embryo-Level Diagnostic Performance Measures | 1-2 Months
  The specificity was calculated for morphology alone prediction and compared to the specificity for adjunct prediction. Comparable calculations was done for sensitivity, negative predictive value, positive predictive value, negative likelihood ratio and positive likelihood ratio. The above measures were given both as an overall and for each panelist, assessing the performance measures without and with adjunct prediction.
Top 2 Embryo Analysis | 1-2 Months
  This analysis included the top 2 embryos selected by each panelist based on morphology alone. The assessment of whether or not the OR is significantly greater than 1, was done by the use of a generalized linear mixed model (GLMM)
Treatment Level Analyses | 1-2 Months
  For the performance assessments of treatment level analyses the predicted blastocyst outcome were compared with the actual blastocyst outcome with each treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Belinda Dueholm, MSc, Principal Investigator — Vitrolife A/S
Locations (6):
- United States (6):
  - Fertility Specialists Medical Group, Inc, San Diego, California
  - Laurel Fertility Care, San Francisco, California
  - Pacific Fertility, San Francisco, California
  - South Florida Institute Fro Reproductive Medicine, Miami, Florida
  - Midwest Fertility Institute, Carmel, Indiana
  - New York Fertility Institute, New York, New York

IPD SHARING:
Plan to Share IPD: No
Patient data are confidential

REFERENCES:
- [Result] Petersen BM, Boel M, Montag M, Gardner DK. Development of a generally applicable morphokinetic algorithm capable of predicting the implantation potential of embryos transferred on Day 3. Hum Reprod. 2016 Oct;31(10):2231-44. doi: 10.1093/humrep/dew188. Epub 2016 Sep 8. PMID 27609980